CLINICAL TRIAL: NCT00779467
Title: Epidural Neostigmine Dose Response for the Treatment of Labor Pain
Brief Title: Epidural Neostigmine for Labor Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00005917
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Labor Pain
Keywords: non narcotic; epidural; labor pain; Non narcotic treatment of labor pain
MeSH Terms: conditions — Labor Pain | interventions — Neostigmine; Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bupivacaine with Neostimgine 8 mcg/ml (Experimental): STUDY DRUG INFUSION WITH NEOSTIGMINE 8 MCG/ML
  Interventions: Drug: Neostigmine; Drug: Bupivacaine
- Bupivacaine and Neostigmine 4 mcg/ml (Experimental): STUDY DRUG INFUSION CONC NEOSTIGMINE 4 MCG/ML
  Interventions: Drug: Neostigmine; Drug: Bupivacaine
- Bupivacaine with Neostigmine 2 mcg/ml (Experimental): STUDY DRUG INFUSION NEOSTIGMINE 2 MCG/ML
  Interventions: Drug: Neostigmine; Drug: Bupivacaine
- BUPIVACAINE WITH FENTANYL 2 MCG/ML (Active Comparator): Bupivacaine with fentanyl 2 mcg/ml. STANDARD INFUSION
  Interventions: Drug: Bupivacaine; Drug: fentanyl

INTERVENTIONS:
Drug: Neostigmine — utilizing 3 different dosages of neostigmine and comparing it to the standard of fentanyl. Infusion runs via PCA throughout labor analgesia.
  Arms: Bupivacaine and Neostigmine 4 mcg/ml; Bupivacaine with Neostigmine 2 mcg/ml; Bupivacaine with Neostimgine 8 mcg/ml
Drug: Bupivacaine
Drug: fentanyl — fentanyl 2 mcg/ml
  Arms: BUPIVACAINE WITH FENTANYL 2 MCG/ML

SUMMARY:
The purpose of this study is to see which dose of epidural neostigmine is the best additive to use with the numbing medication used in an epidural during labor.

DETAILED DESCRIPTION:
This study is examining the use of the non-narcotic medication, neostigmine, in combination with the local anesthetic bupivacaine when compared with the commonly used narcotic fentanyl in providing pain relief with the fewest side effects in labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy
* Term pregnancy ( > 37 weeks)
* Primiparous or multiparous
* Induction or spontaneous labor greater or = 18 years of age
* Cervical exam on entry </=5 cm

Exclusion Criteria:

* Weight > 115 kg
* Non-English speaking
* IV analgesics within 60 minutes prior to epidural being administered
* Allergy to local anesthetics or neostigmine

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Pan, MD, Principal Investigator — Wake Forest University Health Sciences OB Anesthesia
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine With Neostimgine 8 mcg/ml: STUDY DRUG INFUSION WITH NEOSTIGMINE 8 MCG/ML
  Neostigmine: utilizing 3 different dosages of neostigmine and comparing it to the standard of fentanyl. Infusion runs via PCA throughout labor analgesia.
  Bupivacaine
- Bupivacaine and Neostigmine 4 mcg/ml: STUDY DRUG INFUSION CONC NEOSTIGMINE 4 MCG/ML
  Neostigmine: utilizing 3 different dosages of neostigmine and comparing it to the standard of fentanyl. Infusion runs via PCA throughout labor analgesia.
  Bupivacaine
- Bupivacaine With Neostigmine 2 mcg/ml: STUDY DRUG INFUSION NEOSTIGMINE 2 MCG/ML
  Neostigmine: utilizing 3 different dosages of neostigmine and comparing it to the standard of fentanyl. Infusion runs via PCA throughout labor analgesia.
  Bupivacaine
- BUPIVACAINE WITH FENTANYL 2 MCG/ML: Bupivacaine with fentanyl 2 mcg/ml. STANDARD INFUSION
  Bupivacaine
  fentanyl: fentanyl 2 mcg/ml
Period: Overall Study
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Started | 53 | 45 | 48 | 54
Completed | 38 | 40 | 38 | 35
Not Completed | 15 | 5 | 10 | 19
Not completed — Lack of Efficacy | 11 | 2 | 6 | 11
Not completed — failed inclusion criteria | 3 | 3 | 1 | 2
Not completed — missing data | 1 | 0 | 1 | 4
Not completed — technical issue | 0 | 0 | 2 | 1
Not completed — unavailable research staff | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML | Total
Number analyzed (Participants) | 38 | 40 | 38 | 35 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (5) | 27 (6) | 28 (6) | 27 (6) | 27.5 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 38 | 35 | 151
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Amount of Drug Consumed Per Hour in Each Group(Arm)
Description: Median hourly total bupivacaine consumption. Drug amount consumed per hour of each group (arm)
Time Frame: until delivery
Population: median hourly total bupivacaine consumption in each group, in ml/hr
Measure: Median (Inter-Quartile Range); unit: milliliters per hour
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
milliliters per hour | 16.2 [12 to 23] | 14.6 [12 to 18] | 15.3 [13 to 19] | 16 [13 to 21]

2. Secondary Outcome: Nausea
Description: average maximum nausea score in each group--maternal nausea scored on a 0-no nausea at all up to maximum of 10-worst nausea imaginable
Time Frame: until delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
units on a scale | 1.3 (2.5) | 1.8 (3.0) | 1.8 (3.0) | 1.2 (2.2)

3. Secondary Outcome: Sedation
Description: average maternal sedation score measured on a 0-not sleepy at all up to a maximum of 10-extremely sleepy
Time Frame: until delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
units on a scale | 3.3 (3.0) | 3.4 (3.0) | 3.3 (2.9) | 4.1 (3.0)

4. Secondary Outcome: Shivering
Description: maternal occurrence of shivering--Shivering scored on a 0-no shivering at all up to maximum of 10-shivering uncontrollably
Time Frame: until delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
units on a scale | 0.2 (0.4) | 0.3 (0.4) | 0.3 (0.5) | 0.2 (0.4)

5. Secondary Outcome: Pruritus
Description: the occurrence of pruritis (itching) throughout the labor analgesia infusion--the presence of itching rated on a scale of 0-no itching at all up to a maximum of 10- severe itching.
Time Frame: until delivery
Population: the presence of itching rated on a scale of 0-no itching at all up to a maximum of 10- severe itching.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
units on a scale | 0.05 (0.3) | 0.03 (0.2) | 0.03 (0.2) | 0.9 (1.8)

6. Secondary Outcome: Bromage Score
Description: the incidence of decreased motor block (Bromage score) documented until delivery. Bromage is defined as 0-freely able to move extremities (no motor block) up to 3-unable to move legs or feet (complete motor block)
Time Frame: until delivery
Population: Bromage is defined as 0-freely able to move extremities (no motor block) up to 3-unable to move legs or feet (complete motor block)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
units on a scale | 0.7 (0.7) | 1.1 (1.4) | 1.0 (0.9) | 0.9 (1.3)

7. Secondary Outcome: Patient Satisfaction Scores
Description: maternal reported satisfaction scores of labor analgesia on a scale of 1-5, with 1-not satisfied at all up to 5 -completely satisfied with labor analgesia
Time Frame: within 24 hours post delivery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
units on a scale | 4.5 [3.0 to 5.0] | 4.0 [4.0 to 5.0] | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 5.0]

8. Secondary Outcome: Cesarean Delivery
Description: percentage of subjects in each group requiring a ceserean delivery
Time Frame: occurence
Measure: Number; unit: percentage of subjects in each group
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Number analyzed (Participants) | 38 | 40 | 38 | 35
percentage of subjects in each group | 21 | 15 | 24 | 14

ADVERSE EVENTS:
Arm/Group | Bupivacaine With Neostimgine 8 mcg/ml | Bupivacaine and Neostigmine 4 mcg/ml | Bupivacaine With Neostigmine 2 mcg/ml | BUPIVACAINE WITH FENTANYL 2 MCG/ML
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/38 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes